CLINICAL TRIAL: NCT02941276
Title: Long-term Evaluation of the Effectiveness Of a Novel Intra-oral Electro-stimulator for the Treatment of raDiotherapy-ASsociated Dry Mouth
Brief Title: A Trial Looking at Treating Dry Mouth After Radiotherapy for Head and Neck Cancer
Acronym: LEONIDAS-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11/0138
Record Dates: First submitted 2016-10-12; First posted 2016-10-21 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Xerostomia; Head and Neck Neoplasms
MeSH Terms: conditions — Xerostomia; Head and Neck Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Active electrostimulator device (intra-oral active second generation Saliwell GenNarino) (Saliwell Ltd., Harutzim, Israel)
  Interventions: Device: Active Electrostimulator device
- Group B (Sham Comparator): Sham electrostimulator device (intra-oral sham second generation Saliwell GenNarino) (Saliwell Ltd., Harutzim, Israel)
  Interventions: Device: Sham Electrostimulator device

INTERVENTIONS:
Device: Active Electrostimulator device — Patients who will receive a fully functioning device
  Arms: Group A
Device: Sham Electrostimulator device — Patients who will receive a device that does not release electric stimuli (but provided mechanical/tactile stimulation)
  Arms: Group B

SUMMARY:
This trial is looking at using an intra-oral electrostimulating device for the management of radiotherapy-induced dry mouth.

DETAILED DESCRIPTION:
Dry mouth is a common complaint of radiotherapy for cancer of the head and neck region. It is a distressing often persistent condition which can lead to longlasting oral discomfort, dental infections, diminished quality of life, social isolation and loneliness. Unfortunately, current therapies of dry mouth are often unsatisfactory, expensive and may result in adverse effects. A novel intraoral electronic device has recently been developed to treat dry mouth. The device, acting as a "salivary pacemaker", harmlessly stimulates nerves of the salivary glands and does not cause adverse side effects. The aim of this proposal is to assess the longterm effects of such a device in this population, which have yet to be investigated, to demonstrate whether its daily application is an effective method of lessening dry mouth and improving life quality. 84 individuals will be enrolled in the study to use the device for 12 months, after receiving appropriate instructions. 42 participants (out of 84) will act as controls as they will receive a sham device that will not deliver electric stimuli but only tactile stimulation (like using a chewing gum). All participants will be allowed to continue using their routine local therapy for dry mouth (e.g. artificial saliva) during the study. Each participant will keep a diary relevant to the frequency of use and potential changes in dry mouth sensation. Participants will also be asked to attend hospital appointments to measure changes in saliva production and complete questionnaires on their dry mouth and quality of life. The device has the potential to radically change current clinical practice. If the trial is successful, the use of the device will provide patients having radiation-induced dry mouth with a safe and drug-free therapeutic modality.

ELIGIBILITY:
Inclusion Criteria:

1. To be at least 18 years old
2. To have received more than 40 Gy of external beam RT for cancer in the H&N region at least 4 months before entry into the study
3. To have grade 1 or 2 of RTOG/EORTC Late Radiation Morbidity Scoring Schema
4. To have a degree of minimum degree of dryness of 50mm (≥50mm) on a 100mm VAS scale (0=no dryness; 100

   =maximum dryness).
5. To have demonstrable residual salivary gland function (increase in salivary flow on appropriate stimulation (e.g. chewing paraffin wax)
6. To have at least one parotid gland

Exclusion Criteria:

1. To have severe uncontrolled systemic disease (on the basis of the classification of the American Society of Anesthesiology: ASA IV and ASA V)
2. To have known allergy to materials similar to those used in the investigational product
3. To wear other active implants such as cardiac pacemaker or defibrillator, or hearing aids
4. To have an unstimulated whole salivary flow of 0ml/15min (complete absence of unstimulated salivary flow as measured via sialometry for 15 minutes).
5. To use of pilocarpine as systemic therapy
6. To have grade 3 RTOG/EROTC or no resting saliva (sialometry = 0mL/1.5 min)
7. To have no parotid glands

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2011-11; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Improvement of subjective perception of dry mouth as measured on the Visual Analog Scale | 12 month
  The primary outcome is defined as the proportion of patients reporting a 30% reduction of xerostomia symptoms as evaluated through a 100mm VAS (100mm=maximum dryness).

SECONDARY OUTCOMES:
Salivary function | 12 month
  Improvement of objective salivary function as measured through 5-minutes sialometry
Head and Neck cancer Quality of Life | 12 month
  Improvement in head and neck quality of life as measured on the EORTC QLQ-H&N35
Oral Health Quality of Life | 12 month
  Improvement in oral health quality of life as measured on the OH-QoL16 questionnaire
General quality of Life | 12 month
  Improvement in general quality of life as measured on the SF-36 questionnaire
Participant compliance | 12 month
  Evaluation of patients' tolerance in using the device by using a diary to record daily measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Stefano Fedele, PhD, Principal Investigator — University College, London

IPD SHARING:
Plan to Share IPD: No